CLINICAL TRIAL: NCT02327169
Title: A Multiarm, Open-label, Phase 1b Study of MLN2480 (an Oral A-, B-, and CRAF Inhibitor) in Combination With MLN0128 (an Oral mTORC 1/2 Inhibitor), or Alisertib (an Oral Aurora A Kinase Inhibitor), or Paclitaxel, or Cetuximab, or Irinotecan, in Adult Patients With Advanced Nonhematologic Malignancies
Brief Title: A Study MLN2480 in Combination With MLN0128 or Alisertib, or Paclitaxel, or Cetuximab, or Irinotecan in Adult Participants With Advanced Nonhematologic Malignancies
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Organization: Takeda (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: C28002; 2014-003340-12 (EudraCT Number); U1111-1159-5831 (Other: World Health Organization)
Record Dates: First submitted 2014-12-23; First posted 2014-12-30 (Estimated); Results first posted 2020-02-25 (Actual); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Advanced Nonhematologic Malignancies
Keywords: Drug therapy
MeSH Terms: interventions — tovorafenib; sapanisertib; MLN 8237; Paclitaxel; Cetuximab; Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- MLN2480 + MLN0128 (Experimental): Dose Escalation Phase: MLN2480 100 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and MLN0128 2 mg, capsules, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles.
  Interventions: Drug: MLN2480; Drug: MLN0128
- MLN2480 + Alisertib (Experimental): Dose Escalation Phase: MLN2480 100-200 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and alisertib 30-40 mg, tablets, orally, twice daily (BID) on protocol specified days of a 28-day cycle for up to 12 cycles. The doses of MLN2480 and alisertib were modified during this phase based on tolerability during each 28-day cycle.
  Interventions: Drug: MLN2480; Drug: Alisertib
- MLN2480 + Paclitaxel (Experimental): Dose Escalation Phase: MLN2480 100-200 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 milligram per square meter (mg/m^2), intravenous (IV) infusion, once weekly (QW) for 3 weeks in each 28-day cycle for up to 12 cycles or MLN2480 400-600 mg tablets, orally, QW on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, QW for 3 weeks in each 28-day cycle for up to 12 cycles The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
  Interventions: Drug: MLN2480; Drug: Paclitaxel
- MLN2480 + Cetuximab (Experimental): Dose Escalation Phase: MLN2480 400-600 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and cetuximab administered intravenously at a loading dose of 400 mg/m^2 (cycle 1 Day 1), then at 250 mg/m^2 QW on Days 8, 15, and 22 of cycle 1 and Days 1, 8, 15, and 22 in each additional 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in cetuximab dose was based on the standard of care.
  Interventions: Drug: MLN2480; Drug: Cetuximab
- ML2480 + Irinotecan (Experimental): Dose Escalation Phase: MLN2480 400-600 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and irinotecan 180 mg/m^2, IV infusion over 90 minutes, every other week (Q2W) for 2 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in irinotecan dose was based on the standard of care.
  Interventions: Drug: MLN2480; Drug: Irinotecan
- MLN2480 600 mg + Paclitaxel 80 mg (Dose Expansion Phase) (Experimental): Dose Expansion Phase: MLN2480 600 mg, tablets, orally, once per week on Days 2, 9, 16 and 23 of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg, capsules, orally, once on 1, 8, and 15 of a 28-day cycle for up to 12 cycles.
  Interventions: Drug: MLN2480

INTERVENTIONS:
Drug: MLN2480 — MLN2480 tablets.
  Other Names: TAK-580
Drug: MLN0128 — MLN0128 capsules.
  Arms: MLN2480 + MLN0128
Drug: Alisertib — Alisertib tablets.
  Arms: MLN2480 + Alisertib
Drug: Paclitaxel — Paclitaxel IV infusion.
  Arms: MLN2480 + Paclitaxel
Drug: Cetuximab — Cetuximab IV infusion.
  Arms: MLN2480 + Cetuximab
Drug: Irinotecan — Irinotecan IV infusion.
  Arms: ML2480 + Irinotecan

SUMMARY:
The primary purpose of this study is to determine the safety profile and the maximum tolerated doses (MTDs)/ potential recommended phase 2 doses (RP2Ds) of the combination treatments of MLN2480 + MLN0128, MLN2480 + alisertib, MLN2480 + paclitaxel, MLN2480 + cetuximab, and MLN2480 + irinotecan in participants with advanced nonhematologic malignancies.

DETAILED DESCRIPTION:
The drug being tested in this study is called MLN2480 (TAK-580). MLN2480 was tested to evaluate side effects and determine the maximum tolerated dose (MTD) and recommended dose for future studies when administered in combination with five other medications. This study was to assess the safety of MLN2480 as well as how it is processed by the body in participants with solid nonhematologic malignancies who have failed standard therapies.

The study was to be conducted in two phases, the dose escalation phase and the dose expansion phase. A total of 71 participants were enrolled in the escalation phase. Participants in this phase were assigned to one of the five treatment groups:

* MLN2480 + MLN0128
* MLN2480 + Alisertib
* MLN2480 + Paclitaxel
* MLN2480 + Cetuximab
* MLN2480 + Irinotecan

Once the MTD for each combination treatment arm was established in the escalation phase, one or more of the combination treatments will be selected for the expansion phase. A total of 10 participants were enrolled in the expansion phase.

This multi-centre trial was be conducted worldwide. The overall time to participate in this study is approximately 14 months. Participants made multiple visits to the clinic including an end of study visit 30 days after last dose of study drug for a follow-up assessment.

ELIGIBILITY:
Inclusion Criteria:

All Treatment Arms:

1. Male or female participants 18 years or older.
2. Participants who, in the opinion of the treating physician, have failed standard therapies and for whom a phase 1 trial is an appropriate option.
3. Radiographically or clinically evaluable tumor. For expansion phase: Tumors must be measurable and of the protocol specified genetic mutational status, where applicable.
4. Recovered (ie, less than or equal to [<=] Grade 1 toxicity) from adverse effects (except alopecia) of prior therapy.
5. Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
6. Expected survival time of at least 3 months in the opinion of the investigator.
7. Block of banked tumor tissue and/or greater than or equal to (>=) 10 unstained slides. Participants who satisfy all other eligibility criteria but do not have banked tissue/slides may be asked to consent to baseline biopsy.
8. Suitable vein access for the study-required blood sampling.
9. Thyroid function tests consistent with stable thyroid function. Note: Participants on a stable dose of thyroid replacement therapy for a suggested minimum of 12 weeks before Cycle 1, Day 1 are eligible.
10. Left ventricular ejection fraction (LVEF) of 50 percent (%) or greater, as measured by echocardiogram (ECHO) or multiple-gated acquisition scan (MUGA), within 28 days before the first dose of MLN2480
11. Female participants who are post-menopausal for at least 1 year, surgically sterile, or agree to practice 2 effective methods of contraception through 120 days (4 months) after the last dose of study drug for participants in Arms 1, 2, and 5, and through 6 months for participants in Arms 3 and 4, or agree to practice true abstinence.
12. Male participants who, even if surgically sterilized, agree to practice effective barrier contraception through 120 days (4 months) after the last dose of study drug for participants in Arms 1, 2, and 5, and through 6 months for participants in Arms 3, and 4, or agree to practice true abstinence.
13. Additional inclusion criteria for arm 3 expansion only (MLN2480 + paclitaxel):

    a. Participants with Kirsten rat sarcoma viral oncogene homolog (KRAS) exon 2 or BRAF non-V600 mutation-positive non-small cell lung cancer (NSCLC) who have received a minimum of 1 but not more than 2 prior cytotoxic-approved regimens.
14. Additional inclusion criteria for arms 4 and 5 expansion only (MLN2480 + cetuximab; MLN2480 + irinotecan):

    1. Participants with CRC who have received a minimum of 1 but not more than 2 prior cytotoxic-approved regimens.

Exclusion Criteria:

All treatment arms:

1. Female participants who are pregnant or currently breastfeeding.
2. History of any serious medical or psychiatric illness that could, in the investigator's opinion, potentially interfere with safe protocol completion.
3. History of uncontrolled brain metastasis unless: previously treated with surgery, whole-brain radiation, or stereotactic radiosurgery; stable disease for >= 60 days without steroid use (or stable steroid dose established for >= 28 days before the first dose of MLN2480).
4. Ongoing seizure disorder or a requirement for antiepileptics.
5. Recent prior therapies, including: chemotherapy and hormonal therapy <= 4 weeks or 4 half lives, whichever occurs first, before administration of study drug; immunotherapy/monoclonal antibody use <= 4 weeks before administration of MLN2480; or radiation therapy <= 3 weeks before administration of study drug.
6. Chronic therapeutic corticosteroid use with the exception of replacement therapy for adrenal insufficiency or corticosteroid inhalers.
7. Known history of human immunodeficiency virus infection, hepatitis B, or hepatitis C; Prior allogeneic bone marrow or organ transplantation, or active condition of chronic immune suppression is not allowed.
8. Concomitant use, or administration <= 14 days before first dose of study drug(s), of clinically significant enzyme inducers.
9. Treatment with gemfibrozil (strong Cytochrome P4502C8 [CYP2C8] inhibitor) within 14 days before the first dose of MLN2480.
10. History of or current illicit drug use, drug abuse, or alcohol abuse.
11. Major surgery within 14 days before the first dose of study drug.
12. Inability to comply with study requirements.
13. Other unspecified reasons that, in the opinion of the investigator or Millennium, make the participant unsuitable for enrollment.
14. Additional exclusion criteria for arms 3, 5, and 6 expansion only (MLN2480 + paclitaxel; MLN2480 + irinotecan; MLN2480 monotherapy):

    a. Prior treatment with rapidly accelerated fibrosarcoma (RAF), extracellular signal-regulated kinases (MEK), or other inhibitors of the mitogen-activated protein kinase (MAPK) pathway.
15. Additional exclusion criteria for arm 2 only (MLN2480 + alisertib):

    a. History of uncontrolled sleep apnea syndrome and other conditions that could result in excessive daytime sleepiness, such as severe chronic obstructive pulmonary disease.
16. Additional exclusion criteria for arm 3 only (MLN2480 + paclitaxel):

    a. Known hypersensitivity to paclitaxel, or its components or other drugs formulated in Cremophor® EL (polyoxyethylated castor oil).
17. Additional exclusion criteria for arm 5 only (MLN2480 + irinotecan):

    1. Use of strong or moderate Cytochrome P4503A (CYP3A) inhibitors <= days of the first dose of irinotecan.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Actual)
Dates: Start 2015-01-14 (Actual); Primary Completion 2018-07-02 (Actual); Study Completion 2018-07-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director Clinical Science, Study Director — Takeda
Locations (14):
- United States (5):
  - Massachusetts General Hospital Cancer Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
- France (3):
  - Institut Bergonie, Bordeaux, Gironde
  - Institut Claudius Regaud-Oncopole, Toulouse, Haute Garonne
  - Institut Gustave Roussy, Villejuif, Val De Marne
- Spain (3):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - START Madrid. Fundacion Jimenez Diaz, Madrid
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
- United Kingdom (3):
  - Sarah Cannon Research Institure UK, London, Greater London
  - The Chrisie, Manchester, Greater Manchester
  - Churchill Hospital, Oxford, Oxfordshire

IPD SHARING:
Plan to Share IPD: Yes
Takeda makes patient-level, de-identified data sets and associated documents available for all interventional studies after applicable marketing approvals and commercial availability have been received (or program is completely terminated), an opportunity for the primary publication of the research and final report development has been allowed, and other criteria have been met as set forth in Takeda's Data Sharing Policy (see www.TakedaClinicalTrials.com for details). To obtain access, researchers must submit a legitimate academic research proposal for adjudication by an independent review panel, who will review the scientific merit of the research and the requestor's qualifications and conflict of interest that can result in potential bias. Once approved, qualified researchers who sign a data sharing agreement are provided access to these data in a secure research environment.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 14 investigative sites in the United States, France, Spain, and United Kingdom from 14 September 2016 to 02 July 2018.
Pre-assignment Details: Participants with a diagnosis of advanced nonhematologic malignancies were enrolled in one of the five arm groups: MLN2480 + MLN0128, MLN2480 + Alisertib, MLN2480 + Paclitaxel, MLN2480 + Cetuximab, MLN2480 + Irinotecan.
Groups:
- MLN2480 100 mg + MLN0128 2 mg: Dose Escalation Phase: MLN2480 100 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and MLN0128 2 mg, capsules, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles.
- MLN2480 100 mg + Alisertib 30 mg: Dose Escalation Phase: MLN2480 100 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and alisertib 30 mg, tablets, orally, twice daily (BID) on protocol specified days of a 28-day cycle for up to 12 cycles. The doses of MLN2480 and alisertib were modified during this phase based on tolerability during each 28-day cycle.
- MLN2480 160 mg + Alisertib 30 mg: Dose Escalation Phase: MLN2480 160 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and alisertib 30 mg, tablets, orally, twice daily (BID) on protocol specified days of a 28-day cycle for up to 12 cycles. The doses of MLN2480 and alisertib were modified during this phase based on tolerability during each 28-day cycle.
- MLN2480 200 mg + Alisertib 30 mg: Dose Escalation Phase: MLN2480 200 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and alisertib 30 mg, tablets, orally, BID on protocol specified days of a 28-day cycle for up to 12 cycles. The doses of MLN2480 and alisertib were modified during this phase based on tolerability during each 28-day cycle.
- MLN2480 100 mg + Alisertib 40 mg: Dose Escalation Phase: MLN2480 100 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and alisertib 40 mg, tablets, orally, BID on protocol specified days of a 28-day cycle for up to 12 cycles. The doses of MLN2480 and alisertib were modified during this phase based on tolerability during each 28-day cycle.
- MLN2480 100 mg + Paclitaxel 80 mg/m^2: Dose Escalation Phase: MLN2480 100 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 milligram per square meter (mg/m^2), intravenous (IV) infusion, once weekly (QW) for 3 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
- MLN2480 160 mg + Paclitaxel 80 mg/m^2: Dose Escalation Phase: MLN2480 160 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, QW for 3 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
- MLN2480 200 mg + Paclitaxel 80 mg/m^2: Dose Escalation Phase: MLN2480 200 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, QW for 3 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
- MLN2480 400 mg + Paclitaxel 80 mg/m^2: Dose Escalation Phase: MLN2480 400 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, QW for 3 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
- MLN2480 600 mg + Paclitaxel 80 mg/m^2: Dose Escalation Phase: MLN2480 600 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, QW for 3 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in paclitaxel dose was based on the standard of care.
- MLN2480 400 mg + Cetuximab 250 mg/m^2: Dose Escalation Phase: MLN2480 400 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and cetuximab administered intravenously at a loading dose of 400 mg/m^2 (cycle 1 Day 1), then at 250 mg/m^2 QW on Days 8, 15, and 22 of cycle 1 and Days 1, 8, 15, and 22 in each additional 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in cetuximab dose was based on the standard of care.
- MLN2480 600 mg + Cetuximab 250 mg/m^2: Dose Escalation Phase: MLN2480 600 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and cetuximab administered intravenously at a loading dose of 400 mg/m^2 (cycle 1 Day 1), then at 250 mg/m^2 QW on Days 8, 15, and 22 of cycle 1 and Days 1, 8, 15, and 22 in each additional 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in cetuximab dose was based on the standard of care.
- ML2480 300 mg + Irinotecan 180 mg/m^2: Dose Escalation Phase: MLN2480 300 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and irinotecan 180 mg/m^2, IV infusion over 90 minutes, every other week (Q2W) for 2 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in irinotecan dose was based on the standard of care.
- ML2480 400 mg + Irinotecan 180 mg/m^2: Dose Escalation Phase: MLN2480 400 mg, tablets, orally, once on protocol specified days of a 28-day cycle for up to 12 cycles, and irinotecan 180 mg/m^2, IV infusion over 90 minutes, every other week (Q2W) for 2 weeks in each 28-day cycle for up to 12 cycles. The dose of MLN2480 was modified during this phase based on tolerability during each 28-day cycle. Any changes in irinotecan dose was based on the standard of care.
- Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2: Dose Expansion Phase: MLN2480 600 mg, tablets, orally, once per week on Days 2, 9, 16 and 23 of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg/m^2, IV infusion, once on 1, 8, and 15 of a 28-day cycle for up to 12 cycles.
Period: Overall Study
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Started | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
Not completed — Progressive Disease | 1 | 3 | 4 | 3 | 4 | 3 | 3 | 3 | 4 | 4 | 4 | 3 | 1 | 3 | 3
Not completed — Adverse Event | 2 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 3 | 0 | 2 | 1
Not completed — Symptomatic Deterioration | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 2 | 1
Not completed — Reason Not Specified | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Not completed — Lost to Follow-up | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population, all participants who received any amount of MLN2480.
Groups:
- Total: Total of all reporting groups
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2 | Total
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10 | 81
Age, Continuous [Mean (Full Range); unit: years] | 57.5 [48 to 61] | 48.0 [37 to 63] | 60.9 [24 to 77] | 51.0 [30 to 64] | 68.0 [59 to 77] | 66.0 [54 to 74] | 60.3 [57 to 65] | 70.0 [62 to 78] | 54.2 [41 to 67] | 65.9 [46 to 77] | 52.8 [37 to 66] | 60.1 [48 to 70] | 62.0 [62 to 62] | 62.3 [46 to 75] | 63.9 [57 to 75] | 62.3 [24 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 3 | 4 | 1 | 6 | 2 | 2 | 3 | 5 | 4 | 2 | 4 | 0 | 3 | 5 | 47
  Male | 1 | 0 | 3 | 2 | 2 | 2 | 1 | 1 | 1 | 4 | 4 | 3 | 1 | 4 | 5 | 34
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Not Hispanic or Latino | 4 | 3 | 7 | 0 | 8 | 3 | 1 | 4 | 5 | 7 | 5 | 4 | 1 | 7 | 6 | 65
  Unknown or Not Reported | 0 | 0 | 0 | 2 | 0 | 1 | 1 | 0 | 1 | 1 | 1 | 3 | 0 | 0 | 4 | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 4 | 3 | 6 | 1 | 8 | 4 | 2 | 4 | 3 | 6 | 6 | 4 | 1 | 7 | 5 | 64
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 2
  Other | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 3
  Not Reported | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 3 | 0 | 0 | 4 | 12
Height [Mean (Full Range); unit: centimetres (cm)] — Population: Number analyzed is the number of participants with data available for height.
  centimetres (cm)
    number analyzed (Participants) | 4 | 3 | 6 | 2 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 5 | 10 | 77
    (all) | 168.9 [158 to 191] | 163.4 [158 to 173] | 166.7 [156 to 175] | 160.3 [158 to 163] | 164.5 [158 to 171] | 167.0 [155 to 178] | 167.7 [161 to 175] | 166.3 [161 to 176] | 159.7 [152 to 168] | 167.3 [147 to 183] | 169.8 [159 to 180] | 167.4 [147 to 180] | 182.5 [182.5 to 182.5] | 172.3 [161 to 182] | 162.7 [154 to 173] | 164.7 [147 to 191]
Weight [Mean (Full Range); unit: kilograms (kg)] — Population: Number analyzed is the number of participants with data available for weight.
  kilograms (kg)
    number analyzed (Participants) | 4 | 3 | 6 | 2 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10 | 79
    (all) | 71.55 [49.5 to 111.8] | 80.53 [68.1 to 96.1] | 84.62 [56.5 to 137.6] | 74.15 [71.0 to 77.3] | 63.59 [44.0 to 79.5] | 86.63 [82.9 to 95.5] | 77.40 [60.1 to 109.1] | 65.45 [48.0 to 81.8] | 67.92 [53.2 to 92.0] | 65.79 [44.7 to 99.0] | 76.22 [55.9 to 90.0] | 71.39 [50.0 to 99.0] | 86.50 [86.5 to 86.5] | 74.97 [60.4 to 95.0] | 67.65 [40.0 to 91.9] | 70.31 [40.0 to 137.6]
Body Surface Area (BSA) [Mean (Full Range); unit: square meters (m^2)] — BSA (m^2) = sqrt [height (cm) x weight (kg) / 3600] Population: Number analyzed is the number of participants with data available for body surface area.
  square meters (m^2)
    number analyzed (Participants) | 4 | 3 | 6 | 2 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 5 | 10 | 77
    (all) | 1.818 [1.50 to 2.43] | 1.906 [1.74 to 2.05] | 1.961 [1.59 to 2.57] | 1.817 [1.77 to 1.87] | 1.698 [1.41 to 1.91] | 2.003 [1.89 to 2.12] | 1.884 [1.67 to 2.30] | 1.732 [1.47 to 2.00] | 1.726 [1.51 to 2.01] | 1.738 [1.37 to 2.22] | 1.893 [1.61 to 2.12] | 1.814 [1.43 to 2.22] | 2.094 [2.094 to 2.094] | 1.925 [1.69 to 2.19] | 1.740 [1.31 to 2.06] | 1.846 [1.31 to 2.57]

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE is defined as any untoward medical occurrence in a participant administered a pharmaceutical product; the untoward medical occurrence does not necessarily have a causal relationship with this treatment. An SAE means any untoward medical occurrence that at any dose results in death, is life-threatening, requires in patient hospitalization or prolongation of an existing hospitalization, results in persistent or significant disability or incapacity, is a congenital anomaly/birth defect or is a medically important event.
Time Frame: From Day 1, Cycle 1 through 30 days after the last dose of study drug (up to 13 months)
Population: Safety population was defined as all participants who received any amount of MLN2480.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
Participants
  AEs | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
  SAEs | 2 | 1 | 5 | 1 | 3 | 1 | 1 | 2 | 3 | 4 | 2 | 3 | 0 | 4 | 7

2. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs)
Description: DLT was defined using National Cancer Institute Common Terminology Criteria for Adverse Events version 4.03 and included: any drug-related hematologic toxicity ≥Grade 4 with the exception of Grade 4 neutropenia <7 days duration; Grade 3 or 4 neutropenia with fever >38.5 degrees Celsius and/or infection or neutropenia requiring colony-stimulating factor OR non-hematologic DLTs that were any Grade 3, 4, or 5 toxicity with the following exceptions: Grade 3 nausea, vomiting, diarrhea, and dehydration occurring in a setting of inadequate treatment; inadequately treated hypersensitivity reactions; Grade 3 elevated transaminases or urine electrolyte abnormality ≤1 week in duration; Grade 3 serum electrolyte abnormality ≤72 hours in duration. DLTs also included: drug-related adverse experience that lead to a dose modification; unresolved drug-related toxicity resulted in delay in initiation of Cycle 2.
Time Frame: From Day 1, Cycle 1 through 30 days after the last dose in Cycle 1 (up to 8 weeks)
Population: The DLT-evaluable population was defined as all participants in the dose escalation phase of the study who either experienced DLT during cycle 1, or completed at least 75% of the scheduled doses in cycle 1 without DLT.
Measure: Count of Participants; unit: Participants
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 8 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
Participants | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 1

3. Primary Outcome: Maximum Tolerated Dose (MTD) for MLN2480
Time Frame: Day 1, Cycle 1 up to 28 days
Population: as for outcome 2
Measure: Number; unit: mg
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 8 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
mg | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | 600 | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established. | NA — MTD was not established.

4. Primary Outcome: Recommended Phase 2 Dose (RP2D) of MLN2480
Time Frame: Day 1, Cycle 1 up to 28 days
Population: as for outcome 2
Measure: Number; unit: mg
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 8 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
mg | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | 600 | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established. | NA — RP2D was not established.

5. Secondary Outcome: Cmax : Maximum Observed Plasma Concentration for MLN2480
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

6. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for MLN0128
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg
Number analyzed (Participants) | 0

7. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Alisertib
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

8. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN2480
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

9. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for MLN0128
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg
Number analyzed (Participants) | 0

10. Secondary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Alisertib
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

11. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for MLN2480
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for MLN0128
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg
Number analyzed (Participants) | 0

13. Secondary Outcome: AUC(0-tau): Area Under the Plasma Concentration-time Curve From Time 0 to Time Tau Over the Dosing Interval for Alisertib
Time Frame: Cycle 1, Day 10 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg
Number analyzed (Participants) | 0 | 0 | 0 | 0

14. Secondary Outcome: Cmax: Maximum Observed Plasma Concentration for Paclitaxel
Time Frame: Cycle 1, Day 15 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Groups:
- Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2: Dose Expansion Phase: MLN2480 600 mg, tablets, orally, once per week on Days 2, 9, 16 and 23 of a 28-day cycle for up to 12 cycles, and paclitaxel 80 mg, capsules, orally, once on 1, 8, and 15 of a 28-day cycle for up to 12 cycles.
Arm/Group | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

15. Secondary Outcome: AUC(0-last): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Paclitaxel
Time Frame: Cycle 1, Day 15 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

16. Secondary Outcome: AUC(0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity, Calculated Using the Observed Value of the Last Quantifiable Concentration for Paclitaxel
Time Frame: Cycle 1, Day 15 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

17. Secondary Outcome: Terminal Elimination Half-life (T1/2) for Paclitaxel
Time Frame: Cycle 1, Day 15 pre-dose and at multiple timepoints (Up to 48 hours) post-dose
Population: The limited PK data did not allow to estimate the PK parameters defined in the protocol.
Arm/Group | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0

18. Secondary Outcome: Objective Response Rate (ORR) Based on Response Evaluation Criteria in Solid Tumors (RECIST)
Description: ORR was defined as the percentage of participants with complete response (CR) or partial response (PR) using Response Evaluation Criteria In Solid Tumors (RECIST) version 1.1. CR: Disappearance of all target lesions, non-target lesions, no new lesions, and normalization of tumor marker level. PR: At least a 30% decrease in the sum of diameters of target lesions, no progression in non-target lesion, and no new lesions.
Time Frame: Baseline then every 2 cycles beginning at Cycle 2, Day 27, until disease progression, death or end of study (Up to 13 months)
Population: Response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at baseline, and 1 postbaseline response assessment.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 1 | 3 | 7 | 3 | 6 | 4 | 3 | 3 | 5 | 6 | 6 | 5 | 1 | 5 | 8
percentage of participants | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 17 [1 to 64] | 75 [19 to 99] | 0 [0 to 0] | 0 [0 to 0] | 40 [5 to 85] | 17 [1 to 64] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 38 [9 to 76]

19. Secondary Outcome: Duration of Response
Description: Duration of Response (DOR) was defined as the time in months from the first documented CR or PR per RECIST v. 1.1 to disease recurrence or disease progression (PD) whichever occurs first.
Time Frame: From first documented response until disease progression (Up to 13 months)
Population: Responders from response-evaluable population was defined as participants who received at least 1 dose of study drug, had measurable disease at baseline, and 1 postbaseline response assessment. For a participant that has not progressed, DOR was censored at the last response assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
months |  |  |  |  | NA [NA to NA] — Median, Lower and upper limits of confidence interval were not estimable due to low number of participants with events. | 3.7 [1.0 to 5.8] |  |  | 6.5 [1.7 to 11.2] | 3.5 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events. |  |  |  |  | 11.5 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events.

20. Secondary Outcome: Time to Response
Description: Time to response was defined as the time in months from the date of first dose of study treatment to the date of the first documentation of a PR or better response.
Time Frame: From date of enrollment to the date of the first documentation of a confirmed response (Up to 13 months)
Population: Response-evaluable population was defined as all participants with measurable disease at baseline who received any amount of MLN2480 and have at least 1 post baseline response assessment.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 1 | 3 | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 3
months |  |  |  |  | 4.2 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events. | 3.7 [2.3 to 3.7] |  |  | 2.7 [1.9 to 3.6] | 1.8 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events. |  |  |  |  | 1.9 [1.9 to 2.0]

21. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS is defined as the time in months from the date of first study drug administration to the date of first documented PD or death due to any cause. PD was based on response evaluation criteria in solid tumors (RECIST V1.1), defined as at least a 20% increase in the sum of diameters of target lesions, taking as reference the smallest sum on study (this includes the baseline sum if that is the smallest on study). In addition to the relative increase of 20%, the sum must also demonstrate an absolute increase of at least 5 mm.
Time Frame: Baseline then every 2 cycles beginning at Cycle 2, Day 27, until disease progression, death or end of study (Approximately up to 13 months)
Population: Safety population is defined as all participants who received any amount of MLN2480. For a participant that has not progressed and has not died, PFS was censored at the last response assessment that is SD or better. Participants with no response assessment were censored at the date of first dose.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
Number analyzed (Participants) | 4 | 3 | 7 | 3 | 8 | 4 | 3 | 4 | 6 | 8 | 6 | 7 | 1 | 7 | 10
months | 0.5 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events. | 1.9 [1.1 to 16.6] | 3.7 [0.4 to 4.6] | 1.9 [1.7 to 4.6] | 9.5 [0.6 to 9.7] | 5.3 [1.3 to 9.5] | 5.5 [1.5 to 7.4] | 2.9 [1.9 to 3.7] | 7.6 [3.6 to 14.7] | 3.3 [1.8 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events. | 2.2 [1.3 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events. | 1.7 [1.0 to 5.4] | 3.6 [NA to NA] — Lower and upper limits of confidence interval were not estimable due to low number of participants with events. | 4.7 [1.8 to NA] — Upper limit of confidence interval was not estimable due to low number of participants with events. | 5.7 [2.2 to 13.3]

ADVERSE EVENTS:
Time Frame: AEs were recorded from the first dose of study drug through 30 days after the last dose of study drug or the start of subsequent antineoplastic therapy, whichever occurred first. SAEs were collected from the signing of Informed Consent through 30 days after the last dose of study drug (Up to 13 months)
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | MLN2480 100 mg + MLN0128 2 mg | MLN2480 100 mg + Alisertib 30 mg | MLN2480 160 mg + Alisertib 30 mg | MLN2480 200 mg + Alisertib 30 mg | MLN2480 100 mg + Alisertib 40 mg | MLN2480 100 mg + Paclitaxel 80 mg/m^2 | MLN2480 160 mg + Paclitaxel 80 mg/m^2 | MLN2480 200 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Paclitaxel 80 mg/m^2 | MLN2480 600 mg + Paclitaxel 80 mg/m^2 | MLN2480 400 mg + Cetuximab 250 mg/m^2 | MLN2480 600 mg + Cetuximab 250 mg/m^2 | ML2480 300 mg + Irinotecan 180 mg/m^2 | ML2480 400 mg + Irinotecan 180 mg/m^2 | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2
All-Cause Mortality (participants affected / at risk) | 0/4 | 0/3 | 2/7 | 0/3 | 1/8 | 0/4 | 0/3 | 0/4 | 0/6 | 0/8 | 2/6 | 2/7 | 0/1 | 0/7 | 2/10
Serious Adverse Events (participants affected / at risk) | 2/4 | 1/3 | 5/7 | 1/3 | 3/8 | 1/4 | 1/3 | 2/4 | 3/6 | 4/8 | 2/6 | 3/7 | 0/1 | 4/7 | 7/10
Other Adverse Events (participants affected / at risk) | 4/4 | 3/3 | 7/7 | 3/3 | 8/8 | 4/4 | 3/3 | 4/4 | 6/6 | 8/8 | 6/6 | 7/7 | 1/1 | 7/7 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | MLN2480 100 mg + MLN0128 2 mg (N=4) | MLN2480 100 mg + Alisertib 30 mg (N=3) | MLN2480 160 mg + Alisertib 30 mg (N=7) | MLN2480 200 mg + Alisertib 30 mg (N=3) | MLN2480 100 mg + Alisertib 40 mg (N=8) | MLN2480 100 mg + Paclitaxel 80 mg/m^2 (N=4) | MLN2480 160 mg + Paclitaxel 80 mg/m^2 (N=3) | MLN2480 200 mg + Paclitaxel 80 mg/m^2 (N=4) | MLN2480 400 mg + Paclitaxel 80 mg/m^2 (N=6) | MLN2480 600 mg + Paclitaxel 80 mg/m^2 (N=8) | MLN2480 400 mg + Cetuximab 250 mg/m^2 (N=6) | MLN2480 600 mg + Cetuximab 250 mg/m^2 (N=7) | ML2480 300 mg + Irinotecan 180 mg/m^2 (N=1) | ML2480 400 mg + Irinotecan 180 mg/m^2 (N=7) | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2 (N=10)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Post-tussive vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Alisertib and was not related.
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Intestinal obstruction (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Alisertib and was not related.
Oesophagitis ulcerative (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN2480 + Paclitaxel in dose expansion phase and was related.
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Sepsis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Alisertib and was not related.
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Cetuximab and was not related.
Gastrointestinal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Cetuximab and was not related.
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Cetuximab and was not related.
Neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 — One treatment-emergent death occurred during treatment with MLN2480 + Cetuximab and was not related.
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 — One treatment-emergent death occurred during treatment with MLN2480 + Paclitaxel in dose expansion phase and was related.
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Metastatic malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0
Neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Splenic haemorrhage (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pyrexia (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
General physical health deterioration (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fluid overload (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | MLN2480 100 mg + MLN0128 2 mg (N=4) | MLN2480 100 mg + Alisertib 30 mg (N=3) | MLN2480 160 mg + Alisertib 30 mg (N=7) | MLN2480 200 mg + Alisertib 30 mg (N=3) | MLN2480 100 mg + Alisertib 40 mg (N=8) | MLN2480 100 mg + Paclitaxel 80 mg/m^2 (N=4) | MLN2480 160 mg + Paclitaxel 80 mg/m^2 (N=3) | MLN2480 200 mg + Paclitaxel 80 mg/m^2 (N=4) | MLN2480 400 mg + Paclitaxel 80 mg/m^2 (N=6) | MLN2480 600 mg + Paclitaxel 80 mg/m^2 (N=8) | MLN2480 400 mg + Cetuximab 250 mg/m^2 (N=6) | MLN2480 600 mg + Cetuximab 250 mg/m^2 (N=7) | ML2480 300 mg + Irinotecan 180 mg/m^2 (N=1) | ML2480 400 mg + Irinotecan 180 mg/m^2 (N=7) | Dose Expansion: MLN2480 600 mg + Paclitaxel 80 mg/m^2 (N=10)
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 6 | 2 | 1 | 0 | 3 | 2 | 4 | 7 | 6 | 4 | 0 | 5 | 6
Decreased appetite (Metabolism and nutrition disorders) | 2 | 1 | 5 | 1 | 5 | 2 | 2 | 1 | 2 | 1 | 0 | 1 | 1 | 2 | 5
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 0 | 1 | 4
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 0 | 2 | 0 | 0 | 2 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 1 | 1 | 4 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 1 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 3 | 0 | 0 | 0 | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0
Hypercholesterolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lactic acidosis (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nausea (Gastrointestinal disorders) | 2 | 1 | 3 | 1 | 3 | 3 | 1 | 3 | 3 | 1 | 0 | 2 | 1 | 4 | 6
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 2 | 0 | 3 | 1 | 1 | 1 | 4 | 3 | 1 | 2 | 0 | 2 | 3
Constipation (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 4 | 2 | 1 | 3 | 2 | 0 | 0 | 3 | 0 | 2 | 3
Vomiting (Gastrointestinal disorders) | 0 | 1 | 2 | 1 | 3 | 2 | 0 | 1 | 2 | 3 | 1 | 1 | 0 | 4 | 4
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 1 | 3 | 1 | 1 | 2 | 1 | 2 | 2
Abdominal distension (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Haematochezia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Mouth ulceration (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gingival bleeding (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rectal haemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Abdominal mass (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Abdominal tenderness (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Anal fistula (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Aphthous ulcer (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faecal vomiting (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gastric haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Glossitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haemorrhoidal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ileus (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Mouth haemorrhage (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Oral pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Proctalgia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue coated (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Toothache (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Fatigue (General disorders) | 3 | 3 | 5 | 1 | 5 | 2 | 2 | 1 | 3 | 3 | 0 | 2 | 1 | 3 | 2
Asthenia (General disorders) | 0 | 0 | 2 | 1 | 1 | 1 | 1 | 1 | 2 | 1 | 1 | 1 | 0 | 4 | 5
Pyrexia (General disorders) | 2 | 1 | 2 | 1 | 3 | 0 | 0 | 0 | 1 | 2 | 0 | 1 | 0 | 2 | 1
Oedema peripheral (General disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 0 | 4 | 1 | 0 | 1 | 0 | 0 | 2
Chills (General disorders) | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1 | 0
Face oedema (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Non-cardiac chest pain (General disorders) | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1
Pain (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0
Catheter site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Localised oedema (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Administration site extravasation (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Catheter site oedema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Early satiety (General disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Inflammation (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion site pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Unevaluable event (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Vaccination site reaction (General disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 1 | 3 | 3 | 1 | 2 | 3 | 1 | 0 | 0 | 1 | 1 | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2 | 0 | 2 | 1 | 1 | 1 | 0 | 3 | 1 | 2 | 2 | 1 | 0 | 0 | 2
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 4 | 0 | 1 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 3 | 1 | 0 | 0 | 0 | 0
Rash papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Actinic keratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dermatitis contact (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ephelides (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hair colour changes (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Keratosis pilaris (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Miliaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nodular rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Onychoclasis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Petechiae (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Pigmentation disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rash erythematous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 2 | 1 | 1 | 5 | 2 | 2 | 0 | 2 | 1 | 0 | 2 | 0 | 2 | 3
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 1 | 3 | 1 | 0 | 0 | 2 | 3 | 0 | 1 | 0 | 2 | 4
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 1 | 1 | 2 | 1 | 2 | 2 | 0 | 1 | 0 | 0 | 2 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1 | 1 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 1
Upper-airway cough syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Rales (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 1 | 0 | 5 | 0 | 5 | 0 | 3 | 3 | 4 | 4 | 0 | 3 | 1 | 5 | 5
Neutropenia (Blood and lymphatic system disorders) | 0 | 1 | 1 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Leukocytosis (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Weight decreased (Investigations) | 1 | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0 | 1 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Transaminases increased (Investigations) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood bilirubin increased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Haemoglobin decreased (Investigations) | 1 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vitamin D decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0
Weight increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0
Adjusted calcium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
International normalised ratio increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0
Blood alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood magnesium decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urea increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Blood urine present (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Breath sounds abnormal (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Lipase increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Platelet count increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prothrombin level decreased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Troponin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
White blood cell count decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
White blood cell count increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 1 | 2 | 2 | 1 | 1 | 0 | 1 | 2 | 1 | 0 | 0 | 0 | 0 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 1 | 1 | 0 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Groin pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Arthropathy (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Clubbing (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Osteopenia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 1 | 1 | 2 | 1 | 0 | 1 | 2 | 3 | 0 | 1 | 0 | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 1
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 4
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 3 | 1 | 0 | 0 | 0 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Aphasia (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Lethargy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ataxia (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperaesthesia (Nervous system disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Memory impairment (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Motor dysfunction (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Neurotoxicity (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Peripheral sensorimotor neuropathy (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Restless legs syndrome (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sciatica (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vocal cord paralysis (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 1 | 0 | 1 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Influenza (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Lung infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Rash pustular (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Breast abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Furuncle (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Gastroenteritis viral (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Laryngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Nail infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Oral fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Paronychia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pyelonephritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Tongue fungal infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypotension (Vascular disorders) | 2 | 0 | 1 | 0 | 1 | 1 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Flushing (Vascular disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0 | 0
Hot flush (Vascular disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Haematoma (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Pallor (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Vena cava thrombosis (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Vision blurred (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 1
Eyelid oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Eye haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Cataract (Eye disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Eye inflammation (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Ocular hyperaemia (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Periorbital oedema (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 1
Palpitations (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial flutter (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial tachycardia (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Left ventricular dysfunction (Cardiac disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Arrhythmia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dysuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Haematuria (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pollakiuria (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal hypertension (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Urinary incontinence (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Urinary tract obstruction (Renal and urinary disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 3 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Confusional state (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Anxiety (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Melanocytic naevus (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Tumour pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Metastases to skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 2 | 0 | 0 | 0
Cholestasis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hepatocellular injury (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Adrenal insufficiency (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypopituitarism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Thyroiditis (Endocrine disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Incision site pain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Infusion related reaction (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Stoma site haemorrhage (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal haemorrhage (Reproductive system and breast disorders) | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Female genital tract fistula (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vaginal discharge (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Vulvovaginal discomfort (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Food allergy (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Sarcoidosis (Immune system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Deafness unilateral (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Device occlusion (Product Issues) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 1 | 0 | 3 | 1 | 2 | 0 | 0 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Malnutrition (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In general, Investigators may publish clinical data after the earlier of (i) publication by the Sponsor or (ii) 12 months following the abandonment, early termination or database lock; provided a copy of the publication provided to Sponsor at least 30 days ahead of publication, the Sponsor's confidential information is removed as may be requested by Sponsor and Investigator defers publication for up to 60 days in the event Sponsor provides notice that it intends to file a patent application.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-08): https://cdn.clinicaltrials.gov/large-docs/69/NCT02327169/Prot_SAP_000.pdf